CLINICAL TRIAL: NCT01603004
Title: A Pilot Study to Identify Potential Molecular Predictors of Response to Novel Therapies in Metastatic Pancreatic Neuroendocrine Tumors
Brief Title: Potential Molecular Predictors of Response to Novel Therapies in Metastatic Pancreatic Neuroendocrine Tumors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-058
Record Dates: First submitted 2012-05-16; First posted 2012-05-21 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Pancreatic Neuroendocrine Cancer
Keywords: MRI; CT; 12-058
MeSH Terms: conditions — Somatostatinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- everolimus, sunitinib or traditional chemotherapy: A total of 30 patients with well differentiated pancreatic NETs who have known liver metastases and who are planned to initiate therapy with either targeted (everolimus or sunitinib) or traditional cytotoxic chemotherapy will be recruited for this study. We plan to recruit approximately 10 patients for each therapy (everolimus, sunitinib, cytotoxic chemotherapy). Evidence of metastatic disease will be determined at the discretion of the oncologist based on available imaging, surgical and pathologic evidence.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Patients will be treated with either sunitinib, everolimus, or traditional chemotherapy according to standard of care. Follow-up with imaging (either MRI or CT) will be performed approximately every 3 months. Unidimensional tumor measurement on standard CT and MRI sequences will be performed, according to guidelines from RECIST v1.1, which will be used to assess for progression of disease. Patients will be followed for up to 5 years. Upon evidence of disease progression, patients will be asked to undergo a post-treatment biopsy. If medically possible and safe, they will stay on the drug until the time of biopsy.

SUMMARY:
Sunitinib and everolimus are two new treatments approved in 2011 for patients with pancreatic neuroendocrine tumors (NETs). In addition, some traditional chemotherapies are often used to treat pancreatic NETs. Traditional chemotherapy is also known as "cytotoxic therapy" and works by killing cells that are actively dividing. There have been no studies to compare the different types of treatment. Since the patient is eligible for treatment with either sunitinib, everolimus or traditional chemotherapy it can help us identify factors that may help future patients benefit from these therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic evidence of well differentiated pancreatic NET
* Evidence of measurable disease by RECIST 1.1. Both patients with synchronous disease and those with prior resected primary cancers will be eligible.
* Patient ≥18 years of age on the day of signing informed consent.
* Planned initiation of active therapy with everolimus ,sunitinib or traditional cytotoxic chemotherapy.

Patients can be included in this study, regardless of prior therapy, but cannot undergo concurrent therapy, such as hepatic artery embolization

* Available archival tissue with adequate FFPE tissue for analysis verified by a pathologist (in cases of biopsies less than 2 cm and/or less than 70% tumor content 10 slides will be required for adequate DNA preparation. For larger biopsies and any resections, 5 slides are sufficient for DNA extraction).

Exclusion Criteria:

* Patient has a history of a second active malignancy with evidence of metastases. Patients with a history of resected prior malignancy are allowed.
* Patient has known psychiatric or substance abuse disorders that would, in the opinion of the treating investigator, interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research patients will be identified by doctors from the Gastrointestinal Oncology Service in the Department of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-05-14 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  standard MRI sequences will be performed, according to guidelines from RECIST 1.1.

SECONDARY OUTCOMES:
Overall survival | 5 years
  standard MRI sequences will be performed, according to guidelines from RECIST 1.1.
best response | 5 years
  standard MRI sequences will be performed, according to guidelines from RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Nitya Raj, M.D, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/